CLINICAL TRIAL: NCT05488457
Title: Pharmacokinetics and Pharmacodynamics of Oxytocin in Cesarean Delivery
Brief Title: Oxytocin Pharmacokinetics and Pharmacodynamics
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB24-0480
Record Dates: First submitted 2022-07-19; First posted 2022-08-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-05

CONDITIONS: Post Partum Hemorrhage; Cesarean Section Complications; Blood Loss
Keywords: Oxytocin; pharmacokinetics and Pharmacodynamics; Uterine Tone; Postpartum; Elective C-Section; Parturients
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage

STUDY DESIGN:
Intervention Model Description: All subjects will receive a 1 IU bolus of deuterated oxytocin (d5OT) intraoperatively during their cesarean delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxytocin PK/PD Arm (Experimental): Eligible subjects will receive a single, 1 IU bolus of deuterated oxytocin (d5OT) intra-operatively, followed by an infusion of standard therapeutic d0 oxytocin immediately after placental delivery.
  Interventions: Drug: deuterated oxytocin (d5OT)

INTERVENTIONS:
Drug: deuterated oxytocin (d5OT) — Subjects will receive a 1 IU bolus of deuterated oxytocin (d5OT) intraoperatively during their nonemergent cesarean delivery.
  Other Names: Deuterium-labeled oxytocin

SUMMARY:
Oxytocin is the first-line drug to promote contraction of the uterus and prevent atony immediately after delivery. Nonetheless, unpredictable uterine atony refractory to oxytocin affects roughly 250,000 parturients annually in the U.S. and rates are increasing. This two-part study will measure the action of oxytocin at cesarean delivery. The first part will measure the pharmacokinetics of a single intravenous (IV) dose of deuterium-labeled oxytocin. The second part will measure the pharmacodynamics of all plasma oxytocin to see how concentrations correspond to the contractile effect on the uterus.

After delivery of the fetus, study subjects will receive a bolus of IV deuterated oxytocin followed by an unlabeled oxytocin infusion. Venous blood samples drawn at multiple time points (within 1 hour after delivery) will be analyzed for plasma concentrations of labeled and unlabeled (endogenous + exogenous infused) oxytocin over time. Plasma concentrations will be compared with 0-10 uterine tone scores measuring uterine contraction strength, to describe the concentration-effect relationship.

The goal of this study is to define both the pharmacokinetics and pharmacodynamics of oxytocin in parturients to help identify the cause(s) of failed first-line oxytocin therapy.

DETAILED DESCRIPTION:
Parturients aged 18-50 with an intrauterine term pregnancy (37 weeks or greater) undergoing non-emergent cesarean delivery at the University of Chicago (UC) and Stanford University will be recruited.

Methods: All subjects will receive standard pre-, intra- and postoperative care for their cesarean delivery with additional study interventions.

Study subjects will have an additional intravenous (IV) catheter inserted for intra-operative study-related blood draws.

A single, 1 International Unit (IU) bolus of deuterated oxytocin (d5OT) will be given to the subject, followed by an infusion of standard protocol oxytocin immediately after placental delivery. IV samples will be drawn from the study IV at 0, 1, 2.5, 5, 10, 20, 30, 45, 60 minutes following administration of the study drug. The samples will be processed, batched and shipped to the central lab being used in this study. Uterine tone scores will be measured simultaneously with blood draws until accurate palpation is no longer possible. Uterine tone score is a 0 to 10 numeric rating scale with 0 to describe unsatisfactory or no uterine tone and 10 to describe perfect uterine tone.

ELIGIBILITY:
Inclusion Criteria

* 18-50 years old
* intrauterine pregnancy
* term (>39 weeks gestation or 37-39 weeks gestation with fetal or maternal medical indication for delivery) pregnancy
* non-emergent (scheduled or unscheduled) cesarean delivery

Exclusion Criteria:

* allergy or contraindication to oxytocin
* inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing non-emergent cesarean delivery
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline plasma concentrations of deuterated oxytocin | Intraoperatively (prior to delivery)
  The plasma concentration of deuterium labelled oxytocin at baseline
Plasma concentrations of deuterated oxytocin at 1 minute | Intraoperatively (1 minute following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 1 minute post-study drug
Plasma concentrations of deuterated oxytocin at 2.5 minutes | Intraoperatively (2.5 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 2.5 minutes post-study drug
Plasma concentrations of deuterated oxytocin at 5 minutes | Intraoperatively (5 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 5 minutes post-study drug
Plasma concentrations of deuterated oxytocin at 10 minutes | Intraoperatively (10 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 10 minutes post-study drug
Plasma concentrations of deuterated oxytocin at 15 minutes | Intraoperatively (15 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 15 minutes post-study drug
Plasma concentrations of deuterated oxytocin at 20 minutes | Intraoperatively (20 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 20 minutes post-study drug
Plasma concentrations of deuterated oxytocin at 30 minutes | Intraoperatively (30 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 30 minutes post-study drug
Plasma concentrations of deuterated oxytocin at 45 minutes | Intraoperatively (45 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 45 minutes post-study drug
Plasma concentrations of deuterated oxytocin at 60 minutes | Intraoperatively (60 minutes following study drug administration)
  The plasma concentration of deuterium labelled oxytocin at 60 minutes post-study drug
0-10 Uterine Tone Score | Intraoperatively (at the time of study drug administration)
  Uterine tone will be ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (1 minute following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (2.5 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (5 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (10 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (15 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (20 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (30 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (45 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.
0-10 Uterine Tone Score | Intraoperatively (60 minutes following study drug administration)
  Uterine tone ranked by the obstetrician on a 0-10 scale by palpation of the uterus. A score of 0 will represent 'no tone' and a score of 10 will represent 'perfect tone'. The relationship between plasma concentrations and clinical effect will be determined for pharmacodynamic modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Naida M Cole, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No